CLINICAL TRIAL: NCT05023707
Title: Pilot Study of the Safety and Efficacy of Anti-FLT3 Chimeric Antigen Receptor Engineered T-Cells in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Anti-FLT3 CAR T-cell Therapy in FLT3 Positive Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Second People's Hospital of Huai'an (Other); PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021136
Record Dates: First submitted 2021-08-10; First posted 2021-08-26 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3,CAR-T,AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T infusion (Experimental): FLT3 positive relapsed or refractory acute myeloid leukemia
  Interventions: Biological: anti-FLT3 CAR-T

INTERVENTIONS:
Biological: anti-FLT3 CAR-T — Single intravenous infusion of anti-FLT3 CAR-T cells

SUMMARY:
This is a prospective,open-label, phase1/2 study to evaluate the safety and efficacy of anti-FLT3 chimeric antigen receptor engineered T cell immunotherapy (CART) in the treatment of FLT3 positive relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
The patients will receive infusion of anti-FLT3 CAR T-cells targeting FLT3 to evaluate the safety and efficacy of anti-FLT3 CAR T-Cells in relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* FLT3 positive relapsed/refractory acute myeloid leukemia
* Age 16-65 years.
* Left ventricular ejection fractions ≥ 0.5 by echocardiography
* Creatinine < 1.5x upper limit of normal.
* Aspartate aminotransferase/aspartate aminotransferase ≤ 2.5x upper limit of normal
* Total bilirubin ≤ 1.5x upper limit of normal
* Karnofsky performance status ≥ 60
* Expected survival time ≥ 3 months (according to investigator's judgement)

Exclusion Criteria:

* Patients are pregnant or lactating
* Uncontrolled active infection
* Grade III/IV cardiovascular disability according to the New York Heart
* Association Classification
* Active hepatitis B or hepatitis C infection
* Patients with HIV infection
* Patients with a history of seizure
* Patients with other contraindications considered unsuitable for participation in this study (according to investigator's judgement)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)：Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)：All CR criteria except for residual neutropenia (<1.0 x 109/L) or thrombocytopenia (<100 x 109/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Event-free survival (EFS) | 2 years
  time from enrollment to the date of primary refractory disease, or relapse from CR or CRi, or death from any cause
Cumulative incidence of relapse(CIR) | 2 years
  time from the date of achievement of a remission until the date of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China